CLINICAL TRIAL: NCT03582241
Title: Retrospective Study of AML Relapses Using Targeted NGS Analysis
Brief Title: NGS in AML Relapse
Acronym: NGSAML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7106
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Relapse; Mutations
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myeloid leukemia (AML) relapse is often associated with a clonal evolution at the cytogenetic and molecular level and therefore represents a challenge in the treatment of AML. Targeted sequencing is now usually done at diagnosis in AML, as only a small core group of genes is frequently mutated in AML and myelodysplastic syndromes. This approach, contrary to WGS is cheaper, together with a rapid turnaround and high sequencing coverage depths allowing the detection of variant allele fractions as low as 2%.

In the investigator's center, targeted analysis of AML patients is routinely realized at diagnosis and at relapse. In thses patients, five different clonal evolution patterns including cytogenetic and molecular analysis at relapse will be evaluated: (1) Stability, defined by no clonal change, (2) Gain, strictly defined by acquisition of additional variations (mutations or cytogenetic alterations), (3) Loss, strictly defined by loss of variants or regression, (4) Gain and Loss, indicating the combination of both Gain and Loss patterns, (5) Emergence, defined by the emergence of alterations that were unrelated to those found at diagnosis.

Karyotype and the mutations of up to 40 AML patients benefited from targeted NGS in the clinical hematology laboratory of the Hopitaux Universitaires de Strasbourg both at the time of the diagnosis of and the relapse will be studied, together with clinical and other biological characteristics.

ELIGIBILITY:
* Inclusion criteria:

  * patients with AML that relapsed studied in the clinical laboratory of hematology of the Hopitaux Universitaires de Strasbourg, France
  * given consentment or non-opposition for retrospective anonymous analysis of clinical and data
* Exclusion criteria:

  * person under tutorship-
  * persons who asked to withdraw from the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with AML that relapsed studied in the clinical laboratory of hematology of the Hopitaux Universitaires de Strasbourg, France
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
overall survival of the different clonal evolution patterns | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie, Strasbourg, France